CLINICAL TRIAL: NCT02883530
Title: Refractory Asthma Stratification Programme (RASP) Bronchoscopy Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Collaborators: Genentech, Inc. (Industry); Queen's University, Belfast (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0568
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Persistent Asthma
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Blood DNA, broncial bipsies and brushings Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Biomarker optimised patients: Optimised biomarker/Th2 low n=40
  Interventions: Procedure: Bronchoscopy
- non -optimised/Th2 low patients: Patients identified in clinic with FeNO <30 ppb. Those who at screening demonstrate FeNO <30 ppb and blood eosinophil count ≤0.20 x109/L will be considered to be non-optimised biomarker-low patients (Th2-low) and will proceed to bronchoscopy n=80
  Interventions: Procedure: Bronchoscopy
- corticosteroid-resistant biomarker: Patients identified in clinic with FeNO >45 ppb who have failed to suppress their FeNO during FeNO suppression testing. These patients are considered adherent to inhaled corticosteroids. Those who at screening also demonstrate blood eosinophils of >0.3x109/L n=40
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Flexible bronchoscopy will be performed under conscious sedation (with premedication using a mild sedative such as 1-2.5 mg IV midazolam) followed by use of topical anaesthesia (lidocaine spray) on the throat, vocal cords, and trachea in order to investigate the airways. The procedure allows sampling of the airway tissue to allow for laboratory analysis. Three brushings of a small area of the epithelial surface of an airway will be performed via a specialised channel of the bronchoscope with the use of a sterile cytology brush and up to eight 2-mm endobronchial biopsies.

SUMMARY:
The Investigators hypothesise that asthma is not a single disease, but a syndrome resulting from several distinct underlying disease processes known as endotypes. There are approximately 30,000 genes in humans, and each gene is responsible for the production of a particular protein. Using a technique called "whole genome expression profiling" The Investigators have undertaken a small study looking at the activity of all 30,000 genes in the airway tissue of people with asthma. This work has identified 3 mutually exclusive distinct molecular patterns (endotypes) of severe asthma and has identified other potentially important molecular targets (manuscripts in preparation). In particular,the Investigators have found that 25-50% of patients have asthma associated with the activity of proteins called Th2 cytokines (Th2-high asthma). New treatments are in development that target this pathway. However, the Investigators do not know what is driving severe asthma in patients who do not express these Th2 cytokines. The aim of this study is to investigate in more detail the molecular mechanisms driving severe asthma in patients who do not express Th2 cytokines (Th2-low asthma), so that the Investigators can identify new targets for treatment in this group. To do this the Investigators will collect airway tissue via a telescope (bronchoscope), and analyse gene and protein expression in the tissue. The Investigators will then compare the molecular activity between patients with Th2-high and Th2-low asthma, and healthy control subjects (data obtained from a parallel study).

DETAILED DESCRIPTION:
Asthma is a very common disorder which causes a great deal of distress for patients, and occasionally results in premature death. Approximately 10% of people with asthma have severe disease which is not helped by current treatments; The Investigators need to find new treatments for these patients urgently. Patients with asthma are not all the same, but have distinct features which characterise their asthma.The Investigators therefore hypothesise that asthma is not a single disease, but a syndrome resulting from several distinct underlying disease processes known as endotypes. There are approximately 30,000 genes in humans, and each gene is responsible for the production of a particular protein. Using a technique called "whole genome expression profiling" The Investigators have undertaken a small study looking at the activity of all 30,000 genes in the airway tissue of people with asthma. This work has identified 3 mutually exclusive distinct molecular patterns (endotypes) of severe asthma and has identified other potentially important molecular targets (manuscripts in preparation).

In particular, the Investigators have found that 25-50% of patients have asthma associated with the activity of proteins called Th2 cytokines (Th2-high asthma). New treatments are in development that target this pathway. However, the Investigators do not know what is driving severe asthma in patients who do not express these Th2 cytokines. The aim of this study is to investigate in more detail the molecular mechanisms driving severe asthma in patients who do not express Th2 cytokines (Th2-low asthma), so that the Investigators can identify new targets for treatment in this group. To do this the Investigators will collect airway tissue via a telescope (bronchoscope), and analyse gene and protein expression in the tissue. The Investigators will then compare the molecular activity between patients with Th2-high and Th2-low asthma, and healthy control subjects (data obtained from a parallel study).

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent and to comply with the study protocol
2. Age 18-65 years at the time of informed consent
3. Severe asthma (BTS treatment step 4/5) despite intensive follow-up by an asthma specialist for at least 3 months
4. Diagnosis of asthma at least 12 months prior to informed consent
5. Baseline post bronchodilator FEV1 ≥ 40% of predicted
6. History of asthma treatment with high doses of inhaled glucocorticosteroids ( ≥1000 μg fluticasone propionate daily or equivalent (Clenil [BDP] 2000 μg, Fostair [BDP] 800 μg, fluticasone furoate 192 μg, budesonide dry powder 1600 μg, ciclesonide 640 μg), and LABA, with or without an additional controller, for at least 3 months prior to screening or previous corticosteroid optimisation (RASP workstrand 1).
7. For patients using oral corticosteroids, adherence with oral prednisolone regimen, as demonstrated by detectable serum prednisolone and evidence of suppressed cortisol within 6 hours of reported daily dose on at least one occasion during the screening period
8. Assessment according to the standards of the BTS UK Difficult Asthma Network or equivalent
9. Chest X-ray or computed tomography (CT) scan obtained within 12 months prior to consent (Visit 1) or chest X-ray during the screening period (prior to Visit 2) confirming the absence of other clinically significant lung disease
10. Documented history of bronchodilator reversibility response of ≥12% and ≥ 200 mL within the past 18 months, as demonstrated by any of the following:

    i) Documented airflow obstruction (FEV1/forced vital capacity [FVC] <70%), where FEV1 has varied by ≥ 12% either spontaneously or in response to oral corticosteroid therapy, or ii) PC20 (provocative concentration of methacholine producing a 20% fall in FEV1) to methacholine <8 mg/mL indicating the presence of airway hyperresponsiveness, or iii) change in FEV1 by ≥ 12% and ≥200 mL after acute reversibility testing with 400 μg albuterol or 2.5-5 mg nebulized salbutamol

    Exclusion Criteria:
    * Treatment with intravenous [IV], intramuscular [IM]) or intraarticular corticosteroids within 4 weeks prior to Visit 1 or during the screening period for any reason, including an acute exacerbation event
    * A severe asthma exacerbation requiring oral corticosteroids within 4 weeks. The patient has had an exacerbation of asthma requiring the new administration of oral steroids or an increase of at least 10 mg in their usual oral prednisolone dose within the last 4 weeks - defined from the last day of adjusted prednisolone therapy (such patients can re-screened >4 weeks from the last exacerbation)..
    * Infection that meets any of the following criteria:

      * Any infection that resulted in hospital admission for ≥24 hours within 4 weeks prior to Visit 1 or during screening
      * Any infection that required treatment with IV or IM antibiotics within 4 weeks prior to Visit 1 or during screening
      * Any active infection that required treatment with oral antibiotics within 2 weeks prior to Visit 1 or during screening
      * Upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening
      * Antibiotics include any antimicrobial therapy used to treat bacterial, fungal, parasitic, viral, or other infections. Antibiotics prescribed for lung infection prophylaxis would also exclude the patient.
    * Active tuberculosis requiring treatment within 12 months prior to Visit 1 Patients who have completed treatment for tuberculosis at least 12 months prior to Visit 1 and have no evidence of recurrent disease are permitted.
    * Known immunodeficiency, including, but not limited to, HIV infection
    * Evidence of acute or chronic hepatitis or known liver cirrhosis
    * AST, ALT, or total bilirubin elevation ≥ 2.0x the upper limit of normal (ULN) during screening
    * Clinically significant abnormality on screening electrocardiogram (ECG) or laboratory tests (haematology, serum chemistry, and urinalysis) that, in the opinion of the investigator, may pose an additional risk of bronchoscopy
    * History of clinically significant lung disease other than asthma
    * Known current malignancy or current evaluation for a potential malignancy
    * Unable to safely undergo elective flexible fiberoptic bronchoscopy because of any one of the following:

      * History of allergic reactions to local anesthetics to be used in the procedure
      * History of a clinically significant clotting abnormality, including on Screening Coagulation Panel
      * History of acute myocardial infarction, unstable angina, or other medical conditions that, in the opinion of the investigator, may make the patient unsuitable for elective bronchoscopy
    * Other clinically significant medical disease that is uncontrolled despite treatment, that is likely, in the opinion of the investigator, to impact the patient's ability to participate in the study
    * Current smoker, former smoker with smoking history of >15 pack-years A current smoker is defined as someone who has smoked at least one cigarette per day (or pipe, cigar, or marijuana) for ≥ 30 days within the 12 months prior to Visit 1. A pack-year is defined as the average number of packs of cigarettes per day times the number of years of smoking.
    * Use of a licensed or investigational monoclonal antibody including anti-IL 13, anti-IL-4/IL-13, omalizumab, anti-IL-5, or anti-IL 17, within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
    * Use of a systemic immunomodulatory or immunosuppressive therapy (other than a monoclonal antibody or corticosteroids [see separate exclusion]) within 3 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
    * Use of other investigational therapy not described above within 4 weeks or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening

      - Patients participating in a clinical trial that has not been unblinded should be assumed to have received the active drug
    * Initiation of or change in allergen immunotherapy within 3 months prior to Visit 1 or during screening
    * Receipt of a live attenuated vaccine within 4 weeks prior to Visit 1 or during screening
    * Pregnant or lactating
    * History of bronchial thermoplasty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refractory asthma patients attending secondary care refractory asthma clinics within the national health services.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-09-26 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Identification of molecular pathways, identified through gene expression analysis of airway biopsy tissue, related to distinct clinical phenotypes of severe asthma. | 4 weeks

SECONDARY OUTCOMES:
Airway cellularity and structure in relation to clinical phenotype of severe asthma | 4 weeks
Airway protein expression in relation to clinical phenotype of severe asthma | 4 weeks
Peripheral blood gene expression in relation to clinical phenotype of severe asthma | 4 weeks
The airway microbiome in relation to molecular pathways and clinical phenotype of severe asthma | 4 weeks
Differentiation of pathways, biomarkers, and heterogeneity between gene expression and pathophysiology in severe asthma | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bradding, MBBS, Principal Investigator — University of Leicester
Locations (8):
- United Kingdom (8):
  - Belfast Health and Social Care, Belfast
  - Heart Of England NHS Foundation Trust, Birmingham
  - Gartnavel General Hospital, Glasgow
  - University Hospitals of Leicester, Leicester
  - University Hospitals of South Manchester NHS foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford Radcliffe Hospitals NHS Trust, Oxford
  - Southampton University Hospitals NHS TRust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khalfaoui L, Symon FA, Couillard S, Hargadon B, Chaudhuri R, Bicknell S, Mansur AH, Shrimanker R, Hinks TSC, Pavord ID, Fowler SJ, Brown V, McGarvey LP, Heaney LG, Austin CD, Howarth PH, Arron JR, Choy DF, Bradding P. Airway remodelling rather than cellular infiltration characterizes both type2 cytokine biomarker-high and -low severe asthma. Allergy. 2022 Oct;77(10):2974-2986. doi: 10.1111/all.15376. Epub 2022 May 25. PMID 35579040
- [Derived] Couillard S, Shrimanker R, Chaudhuri R, Mansur AH, McGarvey LP, Heaney LG, Fowler SJ, Bradding P, Pavord ID, Hinks TSC. Fractional Exhaled Nitric Oxide Nonsuppression Identifies Corticosteroid-Resistant Type 2 Signaling in Severe Asthma. Am J Respir Crit Care Med. 2021 Sep 15;204(6):731-734. doi: 10.1164/rccm.202104-1040LE. No abstract available. PMID 34129808